CLINICAL TRIAL: NCT07270952
Title: Protocol Efficacy of Mouthwashes in Experimental Gingivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Georgios E. Romanos, Professor, Stony Brook University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB2022-00048
Record Dates: First submitted 2025-11-19; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Gingivitis
Keywords: experimental gingivitis; StellaLife; crossover study; Chlorhexidine
MeSH Terms: conditions — Gingivitis | interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: use of StellaLife for 2 weeks in the one arm (17 patients) and then mouth rinse with Chlorhexidine for 2 weeks (the same patients); another group (17 patients) will use first Chlorhexidine and then StellaLife (crossover study)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- StellaLife (Experimental): StellaLife mouthwash for 2 weeks without tooth brushing
  Interventions: Drug: StellaLife
- Chlorhexidine (Experimental)
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: StellaLife — StellaLife will be used in an experimental gingivitis model
  Arms: StellaLife
Drug: Chlorhexidine — Chlorhexidine in 2 different arms in an experimental gingivitis model
  Arms: Chlorhexidine

SUMMARY:
This research was performed to find out the clinical efficacy and the anti-plaque and anti-gingivitis properties of a new oral health product (mouthwash and oral gel; StellaLife) compared to chlorhexidine. This is important since Chlorhexidine (CHX) has side effects, like it alters taste sensation, stains the teeth, and contains alcohol compared to the herbal based StellaLife.

DETAILED DESCRIPTION:
Objectives: To evaluate the clinical efficacy and the anti-plaque and anti-gingivitis properties of a new oral health product (mouthwash and oral gel; StellaLife) compared to chlorhexidine.

Material and Methods: Two different groups of subjects will be selected for this study. All study participants will have a complete periodontal charting at the initial examination visit (screening visit) and prophylaxis visit. Specifically, periodontal charting with plaque assessment (using disclosing agents), probing measurements (in mm), Gingival Index and gingival crevicular fluid (GCF) analysis (in 2 teeth) will be included.

At the first visit an oral test of the saliva using the OralDNALabs will be used to determine the bacterial load and quality. Then, a professional cleaning and polishing of the teeth will be performed.

The subjects of the Group 1 (test) will use initially a mouth rinse 3x/day with StellaLife (test group) for 1-2 min and one minute test gel (with ingredients) at the gingival margin for 1 min. for a total period of 2 weeks. Toothbrushing and flossing will not be allowed by the subjects. Subjects must avoid eating or drinking for 15 min. after the use of the mouthwash and gel. The gel should be applied for 1 min' to ' apply gel evenly using Q-tip at the neck of the teeth (cervico-gingival junction) on both sides of the teeth.

An oral test of the saliva using the OralDNALabs will be used to determine the bacterial load and quality. Then, a professional cleaning and polishing of the teeth will be performed.

Then, patients will continue the study for an additional period of 2 weeks using only Chlorhexidine mouthwash and placebo gel (without ingredients) without tooth brushing. A new test with OralDNALabs with subsequent periodontal charting will be performed and a prophylaxis visit will be included at the end of the study.

The Group 2 (control)-patients will follow similar protocol starting with use of 0.12% Chlorhexidine (Peridex®) 3x/day as mouthwash for (1-2min) and a placebo control gel (without ingredients) for a period of 2 weeks and then the subjects will start using the StellaLife mouthwash and test gel for 2 weeks (crossover study). Also, the subjects must avoid eating or drinking for 15 min. after the use of the mouthwash and gel.

The GCF will be assessed utilizing the Periotron device at the times of periodontal charting to evaluate changes in volume of GCF (from one and the same site of each participant, one posterior tooth in the maxilla and one in the mandible), comparing the baseline, 2-week, and 4- week (final) visit. The same teeth will be used in all evaluation visits for each individual patient.

The professional cleaning will be performed at the end of the study by a certified dental hygienist to achieve low levels of plaque index and gingival index.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients without periodontal disease

Exclusion Criteria:

* no pregnant women or patient with immunocompromised systemic diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth | 4 weeks
  probing pocket depth measurement (in mm)

SECONDARY OUTCOMES:
Gingival crevicular fluid (GCF) volume | 4 weeks
  The measurement will be performed using the Periotron device (every 2 weeks in each group); from one and the same site of each participant, one posterior tooth in the maxilla and one in the mandible

OTHER OUTCOMES:
Saliva analysis of bacteria | 4 weeks
  OralDNALabs test (Direct Diagnostics); determination of periodontal pathogens, such as A.a., P.g. T.d., T.f. and F.n.

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No